CLINICAL TRIAL: NCT03975465
Title: Effects of Expiratory Muscle Strength Training (EMST) on Long-Term Swallowing Dysfunction in Persons With Head and Neck Cancer (HNCA) Post Irradiation (RT)
Brief Title: EMST and Swallowing in Long-Term Survivors of HNCA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accruals
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: Froedtert Hospital (Other); Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Barbara Pauloski, Associate Professor, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRO32538
Record Dates: First submitted 2019-06-01; First posted 2019-06-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Neoplasms; Deglutition Disorders
Keywords: oropharyngeal cancer; laryngeal cancer; swallow; chemoradiation; expiratory muscle strength training; long-term survivor
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders; Oropharyngeal Neoplasms; Laryngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to an 8-week program of either Expiratory Muscle Strength Training (EMST) or Standard Care in order to examine the impact of EMST on swallowing function
Who Masked: Outcomes Assessor
Masking Description: Researchers assessing the outcomes will not know the arm to which the subject was randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expiratory Muscle Strength Training (Experimental): Patients randomized to the EMST arm will use the EMST150 device as packaged, i.e. following package instructions
  Interventions: Behavioral: Expiratory Muscle Strength Training
- Pharyngeal Muscle Strengthening Exercises (Active Comparator): Patients randomized to Standard Care will receive swallowing exercises designed to strengthen muscles that contribute to pharyngeal phase motor events and increase structural range of motion
  Interventions: Behavioral: Pharyngeal Muscle Strengthening Exercises

INTERVENTIONS:
Behavioral: Expiratory Muscle Strength Training — 8 weeks of EMST at 75% maximum expiratory pressure (MEP)
  Arms: Expiratory Muscle Strength Training
Behavioral: Pharyngeal Muscle Strengthening Exercises — 8 weeks of exercises designed to increase pharyngeal muscle strength for swallowing
  Arms: Pharyngeal Muscle Strengthening Exercises

SUMMARY:
This study is a randomized trial examining the impact of expiratory muscle strength training (EMST) on oral intake, swallowing function, and swallow-related quality of life in persons treated for cancer of the head and neck (HNCA) with radiation therapy or chemoradiotherapy (RT/CRT) at least 5 years previously.

DETAILED DESCRIPTION:
Twenty (20) persons treated for cancer of the head and neck (HNCA) with radiation therapy or chemoradiotherapy (RT/CRT) at least 5 years previously will be randomized to an 8-week program of either EMST only and Standard Care only in order to examine the impact of EMST on swallowing function. The EMST program will consist of 5 sets of 5 breaths, 5 days per week for 8 weeks at 75% of maximum expiratory strength. Patients randomized to the EMST group will use the EMST150 (product name) expiratory muscle strength trainer according to package instructions. Standard Care will include swallowing exercises designed to strengthen muscles that contribute to pharyngeal phase motor events and increase structural range of motion. Subjects will be instructed to practice these exercises following a progressive protocol 5 days per week for 8 weeks.

All subjects will be evaluated at baseline and at the completion of their rehabilitation program. Assessment will include measurement of maximum expiratory pressure (MEP), a videofluoroscopic swallow study (VFSS) to objectively document swallow function, administration of swallow-related quality of life (QOL) questionnaires, and documentation of current diet using the International Dysphagia Diet Standardisation Initiative (IDDSI) Drink Levels and Food Levels.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was treated for cancer in the oral cavity, oropharynx, hypopharynx, larynx, or for an unknown primary at least 5 years prior to enrollment. Subjects may have had surgery as long as a minimum dose of 50 Gy of radiation was part of the treatment;
2. Subject must have a current swallow complaint or impairment; these include but are not limited to reduced oral intake, perceived difficulty with bolus transport (e.g. feeling of food sticking in throat); aspiration on various bolus consistencies;
3. Ability to follow directions and engage in a program of rehabilitation

Exclusion Criteria:

1. the subject's swallowing problems are unrelated to treatment for HNCA (e.g. cognitive impairment, history of stroke);
2. the subject presents with contraindications for EMST as specified in the EMST150 package insert unless cleared for participation by the subject's physician. These conditions include untreated hypertension, untreated gastroesophageal reflux diseas, recent stroke, lung disease, and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Level of Oral Intake (number) | 8 weeks
  Change in Food Level and Drink Level on International Dysphagia Diet Standardisation Initiative (IDDSI) scale will be calculated from baseline to post-treatment.
  IDDSI scale rates the level of liquid or food that the person can eat. Scale values range from 0 to 7, with higher values indicating better outcome (greater ability to eat).
Maximum Expiratory Pressure (MEP) cm H20 | 8 weeks
  Change in maximum expiratory pressure level will be calculated from baseline to post-treatment.
Extent of hyoid movement (mm) | 8 weeks
  From Videofluoroscopic Swallow Studies (VFSS), the change in extent of hyoid movement in mm will be determined from baseline to post-treatment.
Upper esophageal sphincter (UES) opening width (mm) | 8 weeks
  From Videofluoroscopic Swallow Studies (VFSS), the change in width of UES opening width in mm will be determined from baseline to post-treatment.
Presence of pharyngeal residue (dichotomous) | 8 weeks
  From Videofluoroscopic Swallow Studies (VFSS), the presence of residue in the pharynx (yes or no) will be determined from baseline to post-treatment.
Penetration-Aspiration Scale rating (number) | 8 weeks
  From Videofluoroscopic Swallow Studies (VFSS), change in the Penetration-Aspiration Scale (PAS) score will be determined from baseline to post-treatment. Penetration-Aspiration Scale is an 8-point ordinal rating scale that rates the depth to which food or liquid invades the airway. Values range from a minimum of 1 to a maximum of 8; higher values represent worse outcome (i.e. greater depth of invasion into the airway)
Timing of Aspiration (category) | 8 weeks
  From Videofluoroscopic Swallow Studies (VFSS), timing of aspiration will be determined from baseline to post-treatment. Timing is identified as a category, either before, during, or after.

OTHER OUTCOMES:
Eating Assessment Tool (EAT-10) (number) | 8 weeks
  Change in score on the EAT-10 will be calculated from baseline to mid-treatment to post-treatment. EAT-10 is an ordinal rating scale with values that range from 0 to 40, with lower score reflecting better function.
M.D. Anderson Dysphagia Inventory (MDADI) (number) | 8 weeks
  Change in scores on the M.D. Anderson Dysphagia Inventory (MDADI) will be calculated from baseline to post-treatment. MDADI consists of four ordinal rating scales with scores ranging from 0 to 100 with higher score reflecting better function.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pauloski, Ph.D., Principal Investigator — University of Wisconsin, Milwaukee
Locations (2):
- United States (2):
  - University of Wisconsin Milwaukee, Milwaukee, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No